CLINICAL TRIAL: NCT00308438
Title: An Open Label Extension Study of the Safety and Efficacy of ALX-0600 in Subjects With Crohn's Disease Who Completed the Pilot Study Protocol CL0600-008
Brief Title: Safety and Efficacy of ALX-0600 in Subjects With Active Crohn's Disease Who Completed Protocol CL0600-008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0600-009
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2006-03-29 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: Crohn Disease; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects in the study dosed at 0.1 mg/kg teduglutide
  Interventions: Drug: Teduglutide (ALX-0600)

INTERVENTIONS:
Drug: Teduglutide (ALX-0600) — 0.1 mg/kg injected subcutaneously daily
  Other Names: teduglutide

SUMMARY:
The purpose of the study is to determine whether an investigational compound, ALX-0600, is safe and effective in treating Crohn's Disease.

DETAILED DESCRIPTION:
The study is sixteen weeks in duration and there are twelve weeks of once-daily injections into your abdomen or thigh. There are a total of five visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed participation in the Pilot Active Crohn's Disease Study.
* Subjects must continue to meet all inclusion criteria for Pilot Active Crohn's Disease Study with the following exceptions:

  * CDAI score greater than 220
  * Stool samples not required
  * C-reactive protein levels are not an exclusion criterion

Exclusion Criteria:

* Subject must continue to meet all exclusion criteria for Pilot Active Crohn's Disease Study with the following exceptions:

  * Participation in a clinical study of an experimental drug or device within 30 days before signing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2005-11-01 (Actual); Study Completion 2006-06-01 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who are in remission (CDAI score less than 150) at week 12 of this study. | 12 weeks after start of study

SECONDARY OUTCOMES:
The percentage of subjects (of those who achieved response in CL0600-008) who, at week 12 of this study, maintain the response they previously achieved. | 12 weeks after study start
The percentage of subjects who did not respond in CL0600-008 who do respond at week 12 in this study | 12 weeks after study start

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (24):
- United States (20):
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Rx Trials, Washington D.C., District of Columbia
  - Clinical Trials Management of Boca Raton, Boca Raton, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Venture Research, North Miami Beach, Florida
  - Pinnacle Trials, Atlanta, Georgia
  - Saint Joseph's Health System, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Long Island Clinical Research Associates, Great Neck, New York
  - Asher Kornbluth, MD, PC, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Atilla Ertan, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - McGuire DVAMC, Richmond, Virginia
  - Dean Foundation Research Center, Madison, Wisconsin
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Center, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences, Halifax, Nova Scotia
  - Life Screening Centres, Toronto, Ontario

REFERENCES:
- [Background] Buchman AL, Katz S, Fang JC, Bernstein CN, Abou-Assi SG; Teduglutide Study Group. Teduglutide, a novel mucosally active analog of glucagon-like peptide-2 (GLP-2) for the treatment of moderate to severe Crohn's disease. Inflamm Bowel Dis. 2010 Jun;16(6):962-73. doi: 10.1002/ibd.21117. PMID 19821509